CLINICAL TRIAL: NCT01159301
Title: A Phase I Study of Sorafenib in Combination With the Histone Deacetylase Inhibitor, Entinostat in Patients With Advanced Cancers
Brief Title: Entinostat and Sorafenib Tosylate in Treating Patients With Advanced or Metastatic Solid Tumors or Refractory or Relapsed Acute Myeloid Leukemia
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2011-01435; NCI-2011-01435 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CDR0000675600; I-165409 (Other: Roswell Park Cancer Institute); 8272 (Other: CTEP)
Record Dates: First submitted 2010-07-08; First posted 2010-07-09 (Estimated); Last update posted 2013-09-19 (Estimated); Status verified 2013-09

CONDITIONS: Adult Acute Basophilic Leukemia; Adult Acute Eosinophilic Leukemia; Adult Acute Megakaryoblastic Leukemia (M7); Adult Acute Minimally Differentiated Myeloid Leukemia (M0); Adult Acute Monoblastic Leukemia (M5a); Adult Acute Monocytic Leukemia (M5b); Adult Acute Myeloblastic Leukemia With Maturation (M2); Adult Acute Myeloblastic Leukemia Without Maturation (M1); Adult Acute Myeloid Leukemia With 11q23 (MLL) Abnormalities; Adult Acute Myeloid Leukemia With Del(5q); Adult Acute Myeloid Leukemia With Inv(16)(p13;q22); Adult Acute Myeloid Leukemia With t(16;16)(p13;q22); Adult Acute Myeloid Leukemia With t(8;21)(q22;q22); Adult Acute Myelomonocytic Leukemia (M4); Adult Erythroleukemia (M6a); Adult Pure Erythroid Leukemia (M6b); Blastic Phase Chronic Myelogenous Leukemia; Recurrent Adult Acute Myeloid Leukemia; Unspecified Adult Solid Tumor, Protocol Specific
MeSH Terms: conditions — Leukemia, Basophilic, Acute; Leukemia, Eosinophilic, Acute; Leukemia, Megakaryoblastic, Acute; Leukemia, Monocytic, Acute; Leukemia, Myeloid, Acute; Congenital Abnormalities; Leukemia, Myelomonocytic, Acute; Leukemia, Erythroblastic, Acute; Blast Crisis | interventions — entinostat; Sorafenib

ARMS (1):
- Treatment (entinostat, sorafenib tosylate) (Experimental): Patients receive oral entinostat once daily on days 1 and 15 and oral sorafenib tosylate twice daily on days 1-28 (days 15-28 only of course 1). Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: entinostat; Drug: sorafenib tosylate; Other: pharmacological study; Other: laboratory biomarker analysis

INTERVENTIONS:
Drug: entinostat — Given orally (PO)
  Other Names: HDAC inhibitor SNDX-275; SNDX-275
Drug: sorafenib tosylate — Given PO
  Other Names: BAY 43-9006; BAY 43-9006 Tosylate Salt; BAY 54-9085; Nexavar; SFN
Other: pharmacological study — Correlative studies
  Other Names: pharmacological studies
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
This phase I trial is studying the side effects and the best dose of entinostat when given together with sorafenib tosylate in treating patients with advanced or metastatic solid tumors or refractory or relapsed acute myeloid leukemia. Entinostat and sorafenib tosylate may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the maximum-tolerated dose of entinostat in combination with sorafenib tosylate in patients with advanced, inoperable, or metastatic solid tumors.

II. To determine the safety and tolerability of this regimen in these patients.

SECONDARY OBJECTIVES:

I. To determine the pharmacokinetic profile of this regimen in patients with refractory/relapsed acute myeloid leukemia (AML).

II. To assess the preliminary anti-tumor activity of this regimen in patients with advanced, inoperable, or metastatic solid tumors or refractory/relapsed AML.

III. To evaluate histone deacetylase (HDAC) inhibition of histone acetylation in leukemia blast cells.

TERTIARY OBJECTIVES (EXPLORATORY):

I. To evaluate the expression of downstream markers of drug activity such as p38, MCL-1, FLT-3, and VEGFR-2 in leukemia blast cells.

II. To evaluate SNDX-induced expression of p21^WAF1/CIP1 in leukemia blast cells.

OUTLINE: This is a multicenter, dose-escalation study of entinostat.

Patients receive oral entinostat once daily on days 1 and 15 and oral sorafenib tosylate twice daily on days 1-28 (days 15-28 only of course 1). Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

Patients in the expansion cohort undergo blood, bone marrow aspiration, or biopsy for pharmacokinetic studies and biomarker analysis.

After completion of study therapy, patients are followed up for up to 24 months.

ELIGIBILITY:
Inclusion Criteria:

* Must meet 1 of the following criteria:

  * Histologically or cytologically confirmed solid tumors (dose-escalation only)

    * Locally advanced, inoperable, or metastatic disease
    * Evaluable or measurable disease
  * Diagnosis of acute myeloid leukemia (AML) for which no other standard therapy, including stem cell transplantation, is expected to result in meaningful clinical response (expansion cohort only)

    * Refractory or relapsed disease
    * Chronic myelogenous leukemia in blast crisis allowed
    * No acute promyelocytic leukemia with t(15;17)
    * Must consent to have fresh tumor, bone marrow aspirate, and biopsy obtained
* No untreated, symptomatic, or unstable brain metastases
* No active CNS involvement for patients with AML
* ECOG performance status 0-1
* ANC ≥ 1,500/mm³ (dose-escalation only)
* Platelet count ≥ 100,000/mm³ (dose-escalation only)
* Hemoglobin ≥ 10 g/dL (dose-escalation only)
* Total bilirubin ≤ 1.5 times upper limit of normal (ULN)
* ALT and AST ≤ 3 times ULN (≤ 5 times ULN for liver metastasis)
* Creatinine clearance ≥ 40 mL/min
* Albumin > 3.0 g/dL
* Plasma phosphorus > lower limit of normal (with supplementation)
* INR ≤ 1.5
* APTT ≤ 1.5 times ULN (if not on anticoagulants)
* Able to swallow oral medications
* ≥ 16 years old (expanded cohort patients recruited at the University of Colorado site)
* Must have tolerated prior sorafenib tosylate (dose: 400 mg twice daily), if applicable
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective double-barrier contraception during the study and for 90 days after completion of study therapy
* No history of cardiac disease, including any of the following:

  * NYHA class II-IV congestive heart failure
  * Active coronary artery disease
  * Prior diagnosis of bradycardia or other cardiac arrhythmia defined as ≥ grade 2 or uncontrolled hypertension
  * Myocardial infarction (MI) within the past 6 months
  * Persistent tachycardia
  * LVEF < 40% by MUGA
  * Second- or third-degree heart block
  * QTc > 490 msec
  * ST-T wave changes consistent with acute MI or acute ischemia
* No clinically active serious infections defined as ≥ grade 2
* No substance abuse, medical, psychological, or social conditions that may, in the opinion of the Investigator, interfere with the patient's participation or evaluation of the study results
* No condition that is unstable or that could jeopardize the safety of the patient and his/her study compliance
* No known HIV infection
* No significant gastrointestinal disorder that, in the opinion of the Investigator, could interfere with the absorption of entinostat and/or sorafenib tosylate including any of the following:

  * Significant, uncontrolled inflammatory bowel disease
  * Abdominal fistula or gastrointestinal perforation within the past 6 months
  * Extensive small bowel resection
  * Requiring tube feeding or parenteral hydration and/or nutrition
* No concurrent immunosuppressive therapies, including high-dose systemic corticosteroids (> 0.5 mg/kg/day prednisone or equivalent) unless used intermittently or as a tapered course for ≤ 4 weeks
* Concurrent hydroxyurea and/or anagrelide allowed
* Concurrent warfarin allowed provided the dose has been stable for the past 2 months and INR has been between 2 and 3
* More than 4 weeks since prior chemotherapy, immunotherapy, or investigational agents (=< 2 weeks for leukemia patients in expansion cohort)
* More than 2 weeks since prior palliative radiotherapy
* More than 4 weeks since major surgery
* More than 2 weeks since minor surgery (e.g., talc pleurodesis, excisional biopsy, etc.)
* Concurrent hormonal therapies (e.g., LHRH antagonists, megestrol, octreotide, calcitonin, etc.) allowed
* No concurrent strong CYP3A4 inducers or inhibitors, including, but not limited to, any of the following:

  * Valproic acid
  * Rifampin
  * Phenobarbital
  * Phenytoin
  * Carbamazepine
  * Ketoconazole
  * Erythromycin
  * Grapefruit
* No other concurrent anticancer therapy including chemotherapy, radiotherapy (including palliative), or immunotherapy (except hydroxyurea in leukemia patients during course 1)
* No other concurrent investigational agents

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2010-06; Primary Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Maximum-tolerated dose as assessed by the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 4.0 | 28 days
Safety as assessed by the NCI CTCAE version 4.0 | Up to 30 days

SECONDARY OUTCOMES:
Pharmacokinetic profile of sorafenib tosylate | At baseline, and at days 15, 16, and 28 of course 1, and day 1 of course 2
Pharmacokinetic profile of entinostat | At baseline and at days 1, 8, 15, 16, and 22
Objective response rate (ORR) based on the best overall response recorded for each patients or according to Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1 | Up to 30 days
  For ORR the 95% confidence interval will be estimated. The 95% confidence interval for percent of patients in each RECIST response category (i.e., CR, PR, SD, and PD) and disease control rate will also be estimated.

CONTACTS AND LOCATIONS:
Overall Officials: Alex Adjei, Principal Investigator — Roswell Park Cancer Institute
Locations (1):
- Roswell Park Cancer Institute, Buffalo, New York, United States